CLINICAL TRIAL: NCT03597256
Title: A Randomized, Multi-center, Evaluator-blinded, No-treatment Controlled Study to Evaluate the Effectiveness and Safety of Restylane Defyne for Correction of Chin Retrusion
Brief Title: Restylane Defyne for Correction of Chin Retrusion
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Galderma R&D (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 43CH1627
Record Dates: First submitted 2018-07-13; First posted 2018-07-24 (Actual); Results first posted 2024-06-12 (Actual); Last update posted 2024-06-12 (Actual); Status verified 2024-05

CONDITIONS: Chin Retrusion
Keywords: Hyaluronic acid; Chin Retrusion

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment Group (Experimental): Single injection and optional touch-up injection with Restylane Defyne in chin
  Interventions: Device: Restylane Defyne
- Control Group (No Intervention): No treatment

INTERVENTIONS:
Device: Restylane Defyne — Intradermal injection
  Arms: Treatment Group

SUMMARY:
This is a randomized, evaluator-blinded, no-treatment controlled study in subjects with Chin Retrusion.

ELIGIBILITY:
Inclusion Criteria:

1. Participated with signed and dated informed consent form.
2. Men or women aged 18 years of age or older of Chinese origin.
3. Subjects who were seeking augmentation therapy for chin retrusion.
4. GCRS score of 1 or 2 as assessed by the Blinded Evaluator

Exclusion Criteria:

1. Known/previous allergy or hypersensitivity to any injectable hyaluronic acid gel.
2. Known/previous allergy or hypersensitivity to local anaesthetics, e.g. lidocaine or other amide-type anaesthetics.
3. History of severe or multiple allergies, manifested by anaphylaxis.
4. Previous facial surgery, or tissue revitalization treatment with laser or light, needling, mesotherapy, radiofrequency, ultrasound, cryotherapy, chemical peeling or dermabrasion below the level of the horizontal line from subnasale within 6 months before treatment.
5. Previous surgery (including aesthetic facial surgical therapy or liposuction), piercing or tattoo in the area to be treated.
6. Previous tissue augmentation therapy or contouring with any permanent (non-biodegradable) or semi-permanent filler, autologous fat, lifting threads or permanent implant below the level of the horizontal line from subnasale.
7. Other condition that was preventing the subject from entering the study in the Investigator's opinion, e.g. subjects not likely to avoid other facial cosmetic treatments, subjects anticipated to be unreliable, unavailable or incapable of understanding the study assessments or having unrealistic expectations of the treatment result.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 148 (Actual)
Dates: Start 2018-10-08 (Actual); Primary Completion 2019-09-24 (Actual); Study Completion 2020-09-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Q-Med AB, Study Director — Galderma R&D
Locations (1):
- Galderma Research Site, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Xie Y, Zhao H, Wu W, Xu J, Li B, Wu S, Chen K, Bromee T, Li Q. Chin Augmentation and Treatment of Chin Retrusion with a Flexible Hyaluronic Acid Filler in Asian Subjects: A Randomized, Controlled, Evaluator-Blinded Study. Aesthetic Plast Surg. 2024 Mar;48(5):1030-1036. doi: 10.1007/s00266-023-03812-2. Epub 2024 Feb 5. PMID 38315229

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 5 sites in China from 08 Oct 2018 to 09 Sep 2020.
Groups:
- Restylane Defyne (Treatment Group): Participants received an initial treatment with maximum 2 milliliter (mL) of Restylane Defyne on Day 1 for chin retrusion and, if other areas of the chin were treated for optimal chin augumentation, another maximum dosage of 2 mL were recommended at each treatment session, i.e., initial treatment or touch-up treatment respectively. An optional touch-up treatment of maximum 2 mL Restylane Defyne were given at 4 weeks after initial treatment if optimal chin augmentation had not been achieved.
- Control (No Treatment Then Restylane Defyne): Participants did not receive treatment at baseline but offered an initial treatment with 2 mL Restylane Defyne at Month 6 follow-up visit after randomization and optional touch-up treatment at 4 Weeks after initial treatment.
Period: Overall Study
Arm/Group | Restylane Defyne (Treatment Group) | Control (No Treatment Then Restylane Defyne)
Started | 111 | 37
Treated | 111 | 34
Completed | 108 | 32
Not Completed | 3 | 5
Not completed — Lost to Follow-up | 3 | 1
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Could not return for treatment | 0 | 1
Not completed — Moved from location | 0 | 1
Not completed — Not accepted the treatment | 0 | 1

BASELINE CHARACTERISTICS:
Population: Full Analysis Set (FAS) included all participants who were treated with Restylane Defyne or randomized to no-treatment group.
Groups:
- Restylane Defyne (Treatment Group): Participants received an initial treatment with maximum 2 mL of Restylane Defyne on Day 1 for chin retrusion and, if other areas of the chin were treated for optimal chin augumentation, another maximum dosage of 2 mL were recommended at each treatment session, i.e., initial treatment or touch-up treatment respectively. An optional touch-up treatment of maximum 2 mL Restylane Defyne were given at 4 weeks after initial treatment if optimal chin augmentation had not been achieved.
- Total: Total of all reporting groups
Arm/Group | Restylane Defyne (Treatment Group) | Control (No Treatment Then Restylane Defyne) | Total
Number analyzed (Participants) | 111 | 37 | 148
Age, Continuous [Mean (Standard Deviation); unit: years] | 33.4 (8.0) | 32.1 (7.1) | 33.0 (7.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 105 | 35 | 140
  Male | 6 | 2 | 8
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Ethnicity: Han Chinese | 109 | 36 | 145
  Ethnicity: Other | 2 | 1 | 3
Blinded Evaluator Galderma Chin Retrusion Scale [Count of Participants; unit: Participants] — Galderma Chin Retrusion Scale (GCRS) is a validated 4-point scale to assesses the chin retrusion from no retrusion (0) to severe retrusion (3) as follows; "0- No retrusion", "1- Mild retrusion", "2- Moderate retrusion", "3- Severe retrusion".
  Participants
    Score 1 | 39 | 9 | 48
    Score 2 | 72 | 28 | 100

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants (Responders) With At Least 1-Point Improvement From Baseline on the GCRS, as Assessed by the Blinded Evaluator at Month 6 ([Baseline Observation Carried Forward] BOCF Method)
Description: GCRS is a validated 4-point scale to assesses the chin retrusion from no retrusion (0) to severe retrusion (3) which was described as follows; "0- No retrusion", "1- Mild retrusion", "2- Moderate retrusion", "3- Severe retrusion". Responder is defined as a participant with an improvement of at least one grade on the GCRS from baseline. Percentage of responders with at least 1-point improvement from baseline on the GCRS, as measured by the blinded evaluator at Month 6 (after last treatment in treatment group, and after randomization in control group). Missing values at Month 6 are imputed using the BOCF method.
Time Frame: At Month 6
Population: FAS population included all participants who were treated with Restylane Defyne or randomized to no-treatment group.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Restylane Defyne (Treatment Group) | Control (No Treatment Then Restylane Defyne)
Number analyzed (Participants) | 111 | 37
Percentage of participants | 81.1 [72.5 to 87.9] | 5.4 [0.7 to 18.2]

2. Secondary Outcome: Percentage of Participants (Responders) With At Least 1-Point Improvement From Baseline on the GCRS as Assessed by the Blinded Evaluator (Observed Cases)
Description: GCRS is a validated 4-point scale to assesses the chin retrusion from no retrusion (0) to severe retrusion (3) which was described as follows; "0- No retrusion", "1- Mild retrusion", "2- Moderate retrusion", "3- Severe retrusion". Responder is defined as a participant with an improvement of at least one grade on the GCRS from baseline. Percentage of responders, defined by at least 1-point improvement from baseline on the GCRS, as measured by the Blinded Evaluator at 3, 6, 9 and 12 months after last treatment in Treatment group, and at 3 months after randomization, as well as 3, 6, 9 and 12 months after last treatment in Control group for observed cases.
Time Frame: Treatment group: At Months 3, 6, 9, and 12 after last treatment, Control group: At Month 3 after randomization and Months 3, 6, 9 and 12 after last treatment
Population: FAS population included all participants who were treated with Restylane Defyne or randomized to no-treatment group. Here, "number of overall participants analyzed" signifies participants who were evaluable for this outcome measure and "number analyzed" signifies participants who were evaluable for specified timepoints.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Restylane Defyne (Treatment Group) | Control (No Treatment Then Restylane Defyne)
Number analyzed (Participants) | 109 | 35
Percentage of participants
  Month 3 (after last treatment): number analyzed (Participants) | 109 | 32
  Month 3 (after last treatment) | 83.5 [75.2 to 89.9] | 78.1 [60.0 to 90.7]
  Month 6 (after last treatment): number analyzed (Participants) | 107 | 33
  Month 6 (after last treatment) | 84.1 [75.8 to 90.5] | 72.7 [54.5 to 86.7]
  Month 9 (after last treatment): number analyzed (Participants) | 106 | 32
  Month 9 (after last treatment) | 71.7 [62.1 to 80.0] | 62.5 [43.7 to 78.9]
  Month 12 (after last treatment): number analyzed (Participants) | 108 | 32
  Month 12 (after last treatment) | 61.1 [51.3 to 70.3] | 68.8 [50.0 to 83.9]
  Month 3 (after randomization): number analyzed (Participants) | 0 | 35
  Month 3 (after randomization) |  | 8.6 [1.8 to 23.1]

3. Secondary Outcome: Percentage of Participants (Responders) With at Least 1-point Improvement From Baseline on the GCRS, as Assessed by the Treating Investigator
Description: GCRS is a validated 4-point scale to assesses the chin retrusion from no retrusion (0) to severe retrusion (3) which was described as follows; "0- No retrusion", "1- Mild retrusion", "2- Moderate retrusion", "3- Severe retrusion". Responder is defined as a participant with an improvement of at least one grade on the GCRS from baseline. Percentage of responders, defined by at least 1-point improvement from baseline on the GCRS, as assessed by the Treating Investigator at week 4, months 3 and 6.
Time Frame: At Week 4 and Months 3, and 6
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Restylane Defyne (Treatment Group) | Control (No Treatment Then Restylane Defyne)
Number analyzed (Participants) | 111 | 36
Percentage of participants
  At Week 4 | 92.8 [86.3 to 96.8] | 0 [0 to 0]
  At Month 3: number analyzed (Participants) | 109 | 35
  At Month 3 | 84.4 [76.2 to 90.6] | 0 [0 to 0]
  At Month 6: number analyzed (Participants) | 107 | 35
  At Month 6 | 80.4 [71.6 to 87.4] | 0 [0 to 0]

ADVERSE EVENTS:
Time Frame: From baseline up to 20 months
Description: Safety population included all participants who were treated with Restylane Defyne or randomized to no-treatment group.
Groups:
- Control (No Treatment): Participants did not receive treatment at baseline and month 6 follow up visit.
- Control (Restylane Defyne): Participants received initial treatment with 2 mL Restylane Defyne at Month 6 follow-up visit after randomization and optional touch-up treatment at 4 Weeks after initial treatment.
Arm/Group | Restylane Defyne (Treatment Group) | Control (No Treatment) | Control (Restylane Defyne)
All-Cause Mortality (participants affected / at risk) | 0/111 | 0/37 | 0/34
Serious Adverse Events (participants affected / at risk) | 2/111 | 1/37 | 1/34
Other Adverse Events (participants affected / at risk) | 19/111 | 4/37 | 5/34
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Restylane Defyne (Treatment Group) (N=111) | Control (No Treatment) (N=37) | Control (Restylane Defyne) (N=34)
Abnormal liver function (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) — Abnormal liver function was unrelated to the injection procedure and/or the study product.
Cervical squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) — Cervical squamous cell carcinoma was unrelated to the injection procedure and/or the study product.
Uterine subserosal leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) — Uterine subserosal leiomyoma was unrelated to the injection procedure and/or the study product.
Lumbar disc herniation (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) — Lumbar disc herniation was unrelated to the product and/or injection procedure.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Restylane Defyne (Treatment Group) (N=111) | Control (No Treatment) (N=37) | Control (Restylane Defyne) (N=34)
Upper respiratory tract infection (Infections and infestations) | 19 (22) | 4 (4) | 5 (6) — Upper respiratory tract infection was not related to the injection procedure and/or the study product.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Initial publication of data from Study must be a multi-centre publication. Any subsequent publication/presentation must be sent to Sponsor for review 60 days before submission for publication/presentation to allow Sponsor to protect patentable inventions/confidential information. Site and Investigator agree to amend proposed publication/presentation, remove such confidential information from it, or postpone submission for a further 60 days/until intellectual property filings take place.

DOCUMENTS (2):
  • Study Protocol (2018-01-15): https://cdn.clinicaltrials.gov/large-docs/56/NCT03597256/Prot_000.pdf
  • Statistical Analysis Plan (2018-08-23): https://cdn.clinicaltrials.gov/large-docs/56/NCT03597256/SAP_001.pdf